CLINICAL TRIAL: NCT00139581
Title: Comparison of Pimecrolimus Cream 1% Twice-Daily to Once-Daily Dosing in the Management of Atopic Dermatitis in Pediatric Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CASM981C2314
Record Dates: First submitted 2005-08-30; First posted 2005-08-31 (Estimated); Last update posted 2008-04-23 (Estimated); Status verified 2008-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis, children, infants, pimecrolimus, bid, od
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Pimecrolimus b.i.d.
  Interventions: Drug: Pimecrolimus
- 2 (Experimental): Pimecrolimus o.d. and placebo o.d.
  Interventions: Drug: Pimecrolimus

INTERVENTIONS:
Drug: Pimecrolimus — Pimecrolimus cream 1 % applied twice daily (b.i.d.)
  Other Names: Elidel b.i.d.
  Arms: 1
Drug: Pimecrolimus — Pimecrolimus cream 1 % applied once daily (o.d.) and placebo applied once daily (o.d.)
  Other Names: Elidel o.d.
  Arms: 2

SUMMARY:
This study is not being conducted in the United States.

To investigate the relative efficacy of pimecrolimus cream 1% applied twice daily (b.i.d.) versus once daily (o.d.) in preventing the progression to disease "relapse".

ELIGIBILITY:
Inclusion criteria - Screening/Run-In Period

* age >= 2 years through age <=17 years of age
* IGA score of 2, 3, or 4 (mild, moderate, or severe AD) affecting >5% TBSA
* outpatients

Exclusion Criteria:Screening/Run-In period

* subjects who applied topical therapy (e.g. tar, topical corticosteroids) within 2 weeks prior to Screening
* subjects who received phototherapy (e.g. UVB, PUVA, Narrow Band) within 4 weeks of Screening
* subjects who received any systemic immunosuppressant
* subjects who received systemic steroids
* females who are pregnant or breast-feeding, or planning to become pregnant during the study
* subjects who are immunocompromised (e.g. lymphoma, AIDS, Wiskott-Aldrich syndrome) or have a history of malignancy (includes basal cell carcinoma, squamous cell carcinoma, melanoma)
* subjects with open skin infections (bacterial, viral or fungal) if at the application site.
* subjects will HSV (common cold sores) are allowed to participate in the study (if not at the application site).
* subjects who have head lice or scabies
* subjects who present with clinical conditions other than AD that may interfere with the evaluation (e.g., generalized erythroderma, acne, Netherton's Syndrome,psoriasis)
* subjects that require systemic therapy for the treatment of atopic dermatitis
* subjects with poor or no clinical response to tacrolimus ointment (Protopic®) or pimecrolimus cream 1%
* subjects who used any experimental or investigational drug or therapy within 6 weeks prior to Screening
* subjects who intend to use experimental or investigational drug therapy during the course of this study
* subjects with known hypersensitivity to pimecrolimus 1% or related drugs (see Investigator's Brochure)
* subjects who are non-compliant with general medical treatment, or are known to miss appointments, or don't intend to comply with the protocol for the duration of the study
* drug abuse, mental dysfunction, or other factors limiting the subject's ability to cooperate fully with study-related procedures
* subjects known to be unreliable or may be unable to complete the study
* any condition or prior/present treatment that would render the subject ineligible for the study

Inclusion criteria - Double-blind Maintenance treatment period

- Achieve complete remission of active disease (no signs or symptoms of AD) without incidence of "relapse" by the end of 6-week Run-In period (may be earlier); or who achieve "disease improvement" (decrease in IGA score by 1 full point confirmed by the investigator) without incidence of relapse at the end of the 6-week Run-In period

Exclusion criteria - Double-blind Maintenance treatment period

* subjects who experienced a "relapse" during the Run-In period
* subjects who applied topical corticosteroids or any alternative or additional therapy for the treatment of AD during the Run-In period
* subjects with active skin infections (bacterial, viral or fungal) except common cold sores (HSV) at the application site
* subjects who failed to record study medication use (and non use) and dosing regimen during the Run-In period
* subjects who failed to apply open label study drug twice daily until "disease remission" or end of the 6 week Run-In period
* subjects who failed to record concomitant medications during the Run-In period
* failure to return open-label study drug (used, partially used, and unused tubes) at the time double-blind study drug is dispensed. In order to avoid medication error, all open label study drug must be returned to the site before starting the Maintenance period

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2004-09; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Time to relapse of atopic dermatitis (defined as the exacerbation of atopic dermatitis to the level where a topical corticosteroid or alternative therapy is required).
Investigators Global Assessment (IGA) and pruritus (itch) assessment of atopic dermatitis at time of suspected relapse

SECONDARY OUTCOMES:
Time to first recurrence of atopic dermatitis
Eczema Area and Severity Index (EASI) and IGA assessments at several time points.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma AG, Study Chair — Novartis Pharmaceuticals
Locations (1):
- This study is not being conducted in the United States, Novartis Pharma AG, Basel, Switzerland